CLINICAL TRIAL: NCT03355339
Title: The Effect of Binasal Occlusion on Balance Following a Concussion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Jacquie van Ierssel, Principle Investigator, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H06-17-20
Record Dates: First submitted 2017-11-09; First posted 2017-11-28 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Concussion Post Syndrome
Keywords: Balance; Dual-task; King-Devick Test; Saccades; Binasal Occlusion
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binasal occlusion (Experimental): Participants will be fitted with glasses covered with occlusive tape from the inner canthi to the nasal border on each lens.
  Interventions: Device: Binasal occlusion
- No binasal occlusion (Active Comparator): Participants will be fitted with non-occluded glasses.
  Interventions: Device: No binasal occlusion

INTERVENTIONS:
Device: Binasal occlusion — Binasal occlusion glasses
  Arms: Binasal occlusion
Device: No binasal occlusion — Non-occluded glasses
  Arms: No binasal occlusion

SUMMARY:
This study evaluates the effect of binasal occlusion (BNO) glasses on balance and eye movement in adults with dizziness after a concussion. Participants will stand on a force plate while rapidly reading a series of numbers both with and without the BNO glasses. It is thought that the BNO glasses will improve both balance and the time to read the numbers.

DETAILED DESCRIPTION:
While most individuals will recover within the first month after concussion, a significant number will continue to experience dizziness, balance problems, cognitive deficits, and vision problems. Single-task measures of static balance may not be sensitive enough, however, to capture mild postural changes still associated with incomplete recovery. Increasingly there is an interest in dual-task paradigms of balance assessment as a more accurate representation of functional postural control associated with activities of daily living and sport participation. Binasal occlusion (BNO) has been proposed as a means of providing visual stabilization to improve postural control in individuals with vision-related balance problems following a concussion.

ELIGIBILITY:
Inclusion Criteria:

Forty adults with persistent symptoms one month or more following a concussion will be recruited for the study. Individuals will be considered eligible if they have been diagnosed with a concussion as defined in the 2016 Berlin consensus statement (McCrory et al., 2017) as a traumatic brain injury induced by biomechanics forces, which was caused by either a direct or indirect blow to the head, face, neck or elsewhere on the body with an impulsive force transmitted to the head, which may or may not have involved loss of consciousness, and included one or more of the following clinical domains:

* Symptoms (e.g. headache, nausea, fatigue, feeling like in a fog, difficulty concentrating or remembering, and/or emotional lability)
* Physical signs (e.g. loss of consciousness, amnesia, neurological deficit);
* Balance impairment (e.g. gait unsteadiness)
* Behavioural changes (e.g. irritability)
* Cognitive impairment (e.g. slowed reaction times)
* Sleep/wake disturbance (e.g. somnolence, drowsiness) Participants must also meet the following inclusion criteria: (1) aged 18-65 years; (2) sustained the concussion 4 or more weeks ago; (3) report persistent dizziness or balance problems not accounted for by a pre-existing musculoskeletal, neurological, or vestibular condition; (4) have normal vision or visual impairments that can be corrected with contact lenses; (5) are proficient in English or French; (6) are able to provide informed consent.

Exclusion Criteria:

* Do not meet criteria stipulated in the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Postural sway | After one month post-injury. Data collection will occur in one single session per participant upon enrolment in the study.
  The primary outcome of interest is the mean medial/lateral and anterior/posterior velocity of centre of pressure, in addition to the 95% ellipse during different conditions of static balance. The minimal clinical difference considered to demonstrate a change in postural sway is 5cm based on previous validation of the Balance TrackS force plate in a concussed population.

SECONDARY OUTCOMES:
Time to completion of the King-Devick Test (KDT) | After one month post-injury. Data collection will occur in one single session per participant upon enrolment in the study.
  The KDT is a vision-based test of rapid number naming speed that acts as a proxy measure for saccadic eye movement. The KDT consists of a demonstration card, plus a series of 3 increasingly more difficult test cards of variably spaced single digit numbers. Following completion of the demonstration card, participants are asked to read each test card from left to right, top to bottom, as quickly as possible without errors. A summary score of the test is recorded as the total time to complete all 3 test cards, measured in seconds. Time to completion for the KDT will be recorded. Any increase in time compared with a control condition, or any uncorrected errors are considered a significant change.
Saccadic eye movement | After one month post-injury. Data collection will occur in one single session per participant upon enrolment in the study.
  Saccadic eye movement will be assessed with a Tobii™ Pro wearable eye tracker. Tobii™ Pro wearable eye tracker uses infrared video-oculography to analyze patterns of eye movement in terms of fixations and saccades. Longer, more complicated visual tasks, such as rapid number naming, require longer processing times. The number of saccades completed during each balance condition will be recorded by the Tobii™ Pro.
Post-concussion symptom score (PCSS) | After one month post-injury. Data collection will occur in one single session per participant upon enrolment in the study.
  The PCSS is a standardized and easily administered 22-item self-report symptom scale that measures the severity of each symptom experienced that day. Symptoms are reported on a 7-point Likert scale, with 0 and 6 representing anchoring points from the absence of symptoms to the presence of severe symptoms. Results are conveyed as the total symptom score and range from 0-132, with a higher score associated with a higher level of symptoms. Total scores demonstrate high internal consistency in a concussion population (α=0.93), with a 6.8 point change (80% CI) associated with a clinical change in symptoms.
Neck Disability Index (NDI) | After one month post-injury. Data collection will occur in one single session per participant upon enrolment in the study.
  The NDI is the most commonly used self-report outcome measure for neck pain. The index is a simple and quickly administered 10-item questionnaire measured on a 6-point Likert scale from 0=no disability to 5 = full disability. Scores range from 0-50, with 50 representing the highest level of disability. Clinically important difference have been reported with a 5-7 point change in score depending on whether the pain was of musculoskeletal or neural origin.
Dizziness Handicap Inventory (DHI) | After one month post-injury. Data collection will occur in one single session per participant upon enrolment in the study.
  The DHI is a self-report measure of disability associated with dizziness. Internal consistency is high for total scores (α = 0.89). The presence of dizziness-related disability is scored as no (0), sometimes (2), or yes (4). Scores range from 0-100, with a higher score reflecting a greater disability associated with dizziness. Cut-off scores exist for mild (16-34), moderate (36-52), and severe (54+) disability, with an 18-point change in score considered clinically meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Sveistrup, PhD, Principal Investigator — University of Ottawa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Broglio SP, Tomporowski PD, Ferrara MS. Balance performance with a cognitive task: a dual-task testing paradigm. Med Sci Sports Exerc. 2005 Apr;37(4):689-95. doi: 10.1249/01.mss.0000159019.14919.09. PMID 15809571
- [Background] Chang JO, Levy SS, Seay SW, Goble DJ. An alternative to the balance error scoring system: using a low-cost balance board to improve the validity/reliability of sports-related concussion balance testing. Clin J Sport Med. 2014 May;24(3):256-62. doi: 10.1097/JSM.0000000000000016. PMID 24284947
- [Background] Ciuffreda KJ, Yadav NK, Ludlam DP. Effect of binasal occlusion (BNO) on the visual-evoked potential (VEP) in mild traumatic brain injury (mTBI). Brain Inj. 2013;27(1):41-7. doi: 10.3109/02699052.2012.700088. Epub 2012 Aug 17. PMID 22900490
- [Background] Ciuffreda KJ, Yadav NK, Ludlam DP. Binasal Occlusion (BNO), Visual Motion Sensitivity (VMS), and the Visually-Evoked Potential (VEP) in mild Traumatic Brain Injury and Traumatic Brain Injury (mTBI/TBI). Brain Sci. 2017 Aug 9;7(8):98. doi: 10.3390/brainsci7080098. PMID 28792441
- [Background] Degani AM, Santos MM, Leonard CT, Rau TF, Patel SA, Mohapatra S, Danna-Dos-Santos A. The effects of mild traumatic brain injury on postural control. Brain Inj. 2017;31(1):49-56. doi: 10.1080/02699052.2016.1225982. Epub 2016 Dec 12. PMID 27936960
- [Background] Galetta KM, Liu M, Leong DF, Ventura RE, Galetta SL, Balcer LJ. The King-Devick test of rapid number naming for concussion detection: meta-analysis and systematic review of the literature. Concussion. 2015 Sep 10;1(2):CNC8. doi: 10.2217/cnc.15.8. eCollection 2016 Mar. PMID 30202552
- [Background] Galetta KM, Morganroth J, Moehringer N, Mueller B, Hasanaj L, Webb N, Civitano C, Cardone DA, Silverio A, Galetta SL, Balcer LJ. Adding Vision to Concussion Testing: A Prospective Study of Sideline Testing in Youth and Collegiate Athletes. J Neuroophthalmol. 2015 Sep;35(3):235-41. doi: 10.1097/WNO.0000000000000226. PMID 25742059
- [Background] Gallop S. A variation on the use of binasal occlusion glasses - a case study. Journal of Behavioural Optometry 9(2): 31-35, 1998.
- [Background] Gallop S. Viewpoint 4 Binasal Occlusion - Immediate , Sustainable Symptomatic Relief. Optometry & Visual Performance 9(2):31-35, 2014.
- [Background] Goble DJ, Manyak KA, Abdenour TE, Rauh MJ, Baweja HS. AN INITIAL EVALUATION OF THE BTRACKS BALANCE PLATE AND SPORTS BALANCE SOFTWARE FOR CONCUSSION DIAGNOSIS. Int J Sports Phys Ther. 2016 Apr;11(2):149-55. PMID 27104048
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Background] Hunt AW, Mah K, Reed N, Engel L, Keightley M. Oculomotor-Based Vision Assessment in Mild Traumatic Brain Injury: A Systematic Review. J Head Trauma Rehabil. 2016 Jul-Aug;31(4):252-61. doi: 10.1097/HTR.0000000000000174. PMID 26291632
- [Background] Kamins J, Bigler E, Covassin T, Henry L, Kemp S, Leddy JJ, Mayer A, McCrea M, Prins M, Schneider KJ, Valovich McLeod TC, Zemek R, Giza CC. What is the physiological time to recovery after concussion? A systematic review. Br J Sports Med. 2017 Jun;51(12):935-940. doi: 10.1136/bjsports-2016-097464. Epub 2017 Apr 28. PMID 28455363
- [Background] Kleffelgaard I, Roe C, Soberg HL, Bergland A. Associations among self-reported balance problems, post-concussion symptoms and performance-based tests: a longitudinal follow-up study. Disabil Rehabil. 2012;34(9):788-94. doi: 10.3109/09638288.2011.619624. Epub 2011 Dec 9. PMID 22149161
- [Background] Lau BC, Kontos AP, Collins MW, Mucha A, Lovell MR. Which on-field signs/symptoms predict protracted recovery from sport-related concussion among high school football players? Am J Sports Med. 2011 Nov;39(11):2311-8. doi: 10.1177/0363546511410655. Epub 2011 Jun 28. PMID 21712482
- [Background] Levac D, DeMatteo C, Hanna S, Wishart L. Intra-individual variability in recovery from paediatric acquired brain injury: relationship to outcomes at 1 year. Dev Neurorehabil. 2008 Jul;11(3):195-203. doi: 10.1080/17518420802055177. PMID 18608358
- [Background] Lovell MR, Iverson GL, Collins MW, Podell K, Johnston KM, Pardini D, Pardini J, Norwig J, Maroon JC. Measurement of symptoms following sports-related concussion: reliability and normative data for the post-concussion scale. Appl Neuropsychol. 2006;13(3):166-74. doi: 10.1207/s15324826an1303_4. PMID 17361669
- [Background] MacDermid JC, Walton DM, Avery S, Blanchard A, Etruw E, McAlpine C, Goldsmith CH. Measurement properties of the neck disability index: a systematic review. J Orthop Sports Phys Ther. 2009 May;39(5):400-17. doi: 10.2519/jospt.2009.2930. PMID 19521015
- [Background] Marshall S, Bayley M, McCullagh S, Velikonja D, Berrigan L, Ouchterlony D, Weegar K; mTBI Expert Consensus Group. Updated clinical practice guidelines for concussion/mild traumatic brain injury and persistent symptoms. Brain Inj. 2015;29(6):688-700. doi: 10.3109/02699052.2015.1004755. Epub 2015 Apr 14. PMID 25871303
- [Background] Master CL, Scheiman M, Gallaway M, Goodman A, Robinson RL, Master SR, Grady MF. Vision Diagnoses Are Common After Concussion in Adolescents. Clin Pediatr (Phila). 2016 Mar;55(3):260-7. doi: 10.1177/0009922815594367. Epub 2015 Jul 7. PMID 26156977
- [Background] McCrea MA, Nelson LD, Guskiewicz K. Diagnosis and Management of Acute Concussion. Phys Med Rehabil Clin N Am. 2017 May;28(2):271-286. doi: 10.1016/j.pmr.2016.12.005. Epub 2017 Mar 1. PMID 28390513
- [Background] McCrory P, Meeuwisse W, Dvorak J, Aubry M, Bailes J, Broglio S, Cantu RC, Cassidy D, Echemendia RJ, Castellani RJ, Davis GA, Ellenbogen R, Emery C, Engebretsen L, Feddermann-Demont N, Giza CC, Guskiewicz KM, Herring S, Iverson GL, Johnston KM, Kissick J, Kutcher J, Leddy JJ, Maddocks D, Makdissi M, Manley GT, McCrea M, Meehan WP, Nagahiro S, Patricios J, Putukian M, Schneider KJ, Sills A, Tator CH, Turner M, Vos PE. Consensus statement on concussion in sport-the 5th international conference on concussion in sport held in Berlin, October 2016. Br J Sports Med. 2017 Jun;51(11):838-847. doi: 10.1136/bjsports-2017-097699. Epub 2017 Apr 26. No abstract available. PMID 28446457
- [Background] O'Connor SM, Baweja HS, Goble DJ. Validating the BTrackS Balance Plate as a low cost alternative for the measurement of sway-induced center of pressure. J Biomech. 2016 Dec 8;49(16):4142-4145. doi: 10.1016/j.jbiomech.2016.10.020. Epub 2016 Oct 20. PMID 27789036
- [Background] Patricios J, Fuller GW, Ellenbogen R, Herring S, Kutcher JS, Loosemore M, Makdissi M, McCrea M, Putukian M, Schneider KJ. What are the critical elements of sideline screening that can be used to establish the diagnosis of concussion? A systematic review. Br J Sports Med. 2017 Jun;51(11):888-894. doi: 10.1136/bjsports-2016-097441. Epub 2017 Mar 7. PMID 28270437
- [Background] Proctor A. Traumatic brain injury and binasal occlusion. Optometry and Vision Development, 40(1): 45-50, 2009.
- [Background] Rizzo JR, Hudson TE, Dai W, Birkemeier J, Pasculli RM, Selesnick I, Balcer LJ, Galetta SL, Rucker JC. Rapid number naming in chronic concussion: eye movements in the King-Devick test. Ann Clin Transl Neurol. 2016 Sep 1;3(10):801-811. doi: 10.1002/acn3.345. eCollection 2016 Oct. PMID 27752515
- [Background] Rochefort C, Walters-Stewart C, Aglipay M, Barrowman N, Zemek R, Sveistrup H. Balance Markers in Adolescents at 1 Month Postconcussion. Orthop J Sports Med. 2017 Mar 17;5(3):2325967117695507. doi: 10.1177/2325967117695507. eCollection 2017 Mar. PMID 28451603
- [Background] Scoppa F, Capra R, Gallamini M, Shiffer R. Clinical stabilometry standardization: basic definitions--acquisition interval--sampling frequency. Gait Posture. 2013 Feb;37(2):290-2. doi: 10.1016/j.gaitpost.2012.07.009. Epub 2012 Aug 11. PMID 22889928
- [Background] Subotic A, Ting WK, Cusimano MD. Characteristics of the King-Devick test in the assessment of concussed patients in the subacute and later stages after injury. PLoS One. 2017 Aug 31;12(8):e0183092. doi: 10.1371/journal.pone.0183092. eCollection 2017. PMID 28859119
- [Background] Yadav NK, Thiagarajan P, Ciuffreda KJ. Effect of oculomotor vision rehabilitation on the visual-evoked potential and visual attention in mild traumatic brain injury. Brain Inj. 2014;28(7):922-9. doi: 10.3109/02699052.2014.887227. Epub 2014 Feb 24. PMID 24564831
- [Background] Zemek RL, Farion KJ, Sampson M, McGahern C. Prognosticators of persistent symptoms following pediatric concussion: a systematic review. JAMA Pediatr. 2013 Mar 1;167(3):259-65. doi: 10.1001/2013.jamapediatrics.216. PMID 23303474
- See also: Tobii Pro — http://www.tobiipro.com

DOCUMENTS (2):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT03355339/Prot_000.pdf
  • Informed Consent Form (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT03355339/ICF_001.pdf